CLINICAL TRIAL: NCT05143450
Title: The Effect of Applying Manual Pressure Before Vaccination on Pain and Crying Time in Infants
Brief Title: Efficacy of Manual Pressure in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-KAEK-53-21-02
Record Dates: First submitted 2021-11-17; First posted 2021-12-03 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2021-11

CONDITIONS: Pain Management
Keywords: injection; manual pressure; pain; pain management; vaccination
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Before the procedure, manual pressure will be applied to the injection site with the thumb for 10 seconds to the infants by the researcher.
  Interventions: Other: Manual Pressure
- Control Group (No Intervention): No intervention will perform to reduce pain in the control group.

INTERVENTIONS:
Other: Manual Pressure — In the experimental group manual pressure will be applied to the injection site with the thumb for 10 seconds to the infants by the researcher before the procedure. Manual pressure reduces pain within the framework of the gate control theory. According to the gate control theory, when pressure is applied to an area, a fiber transmits the feeling of pressure instead of pain and ultimately the pain sensation is alleviated.
  Arms: Experimental Group

SUMMARY:
Manual pressure is an effective, easy-to-apply, no preparation, and cost-effective method of reducing pain associated with the injection. This study will be carried out to determine the effect of manual pressure applied to the injection site on the pain level and crying time of the infants before the injection of the Diphtheria-Tetanus-Acellular Pertussis Vaccine (DTaP), Inactivated Polio Vaccine (IPV), and Haemophilus Influenzae Type b Vaccine (Hib) (5-in-1) in 2-month-old infants. The study will be conducted with the randomized controlled experimental method. Before the procedure, manual pressure will be applied to the injection site with the thumb for 10 seconds to the infants in the experimental group. No non-pharmacological method will be used before vaccination to the infants in the control group. Pain scores of infants in the intervention and control groups will be evaluated before, during, and after vaccination. In addition, the total crying times of the babies will be calculated and recorded with a stopwatch.

DETAILED DESCRIPTION:
Vaccine injection is one of the most common causes of pain in healthy infants and children. Parents may avoid or delay vaccination to avoid the pain their child experiences repeatedly with vaccination. Avoiding or delaying vaccination by parents may lead to disruption of vaccination programs, and thus an increase in infectious diseases that can be prevented by vaccination. Therefore, the management of pain due to vaccine injection in children is very important. Many non-pharmacological methods are used to control vaccine-related pain in children. Manual pressure, which is one of these methods, is applied to the injection area with the thumb for 10 seconds before the injection. The pain control effect of manual pressure is explained by the gate control theory. According to this theory, the presence and severity of pain depend on the transmission of neurological stimuli. In summary, if the door is open, the warnings reach the level of consciousness and pain is felt, if it is closed, the warnings do not reach the consciousness and pain is not felt. Applications such as rubbing the pain area, pressing with a finger, massage provide closing the door to painful stimuli. The aim of the study is to determine the effect of manual pressure applied to the injection site on the pain level and crying time of the infants before the injection of the DTaP-IPV-Hib vaccine (5-in-1) in 2-month-old infants.The sample size of the study has been determined by the power analysis (G*Power 3.1.9.2), in line with the results obtained from the studies which have been conducted using a similar research method. The sample size was found to be a total of 66 children including minimum of 33 children for each group. It was estimated that case losses may occur and therefore, it was decided to conduct the study with a total of 70 children including 35 children in two groups. Information Form, Face, Legs, Activity, Cry, Consolability (FLACC) Scale, and chronometer will use for data collection. Children's parents who applied to the Kumkapi Family Health Center will be given information about the study. Information about children and their parents included in the study will ask by the researcher through face-to-face interviews and these data will record in 'Information Form' five minutes before the procedure.

Before the procedure, manual pressure will be applied to the injection site with the thumb for 10 seconds to the infants in the experimental group. No non-pharmacological method will be used before vaccination to the infants in the control group. The latero-femoral region (vastus lateralis muscle) will be used as the injection site for vaccination. All infants in the intervention and control groups will be accompanied by their parents throughout the procedure. In addition, the chronometer will be started when the baby starts to cry, and the chronometer will be stopped when the crying stops. Total crying time will be recorded on the Information Form. Before, during, and after vaccination children's pain will evaluate with the FLACC Scale by the healthcare provider who performs the injection. Before and during venipuncture children's pain will evaluate with the FLACC Scale and their emotional status will evaluate with the Children's Emotional Manifestation Scale by the healthcare provider who performs the venipuncture procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy baby born at term
* Being 4 months old
* Having no chronic disease,
* Having no neurological disease.
* Not taking an analgesic drug within 24 hours before vaccination.

Exclusion Criteria:

* Being an unhealthy baby born at preterm or post-term,
* Being younger or older than 4 months old,
* Having a chronic disease,
* Having a neurological disease,
* Taking an analgesic drug within 24 hours before vaccination.

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Change of Pain | Before vaccine injection, when the vaccine starts to be injected and immediately after the injector was removed.
  Pain will assess by the healthcare provider who performs the venipuncture procedure with the FLACC (Face, Legs, Activity, Cry, Consolability) Scale. This scale was developed to evaluate the pain of children aged 2 months to 7 years. The child's facial expression, leg movements, activity, crying, and comfortability behaviors are evaluated in relation to pain. These five behaviors are rated with 0, 1, or 2 points. The total score of the scale ranges from 0 to 10, and a high score indicates that the child has more pain. '0' points from the scale indicate no pain, '1-3' points indicate mild pain, '4-6' points indicate moderate pain, and '7-10' points indicate severe pain.

SECONDARY OUTCOMES:
Crying time | During vaccine injection and immediately after injection
  Crying time throughout vaccine injections will be calculated for each infant using a chronometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Kumkapi Family Health Center, Istanbul, Turkey (Türkiye)